CLINICAL TRIAL: NCT05048095
Title: The Use of AI as a Third Reader and During Consensus in a Double Reading Breast Cancer Screening Program in Sweden
Brief Title: Artificial Intelligence in Breast Cancer Screening in Region Östergötland Linkoping
Acronym: AI-ROL
Status: Completed | Type: Observational
Sponsor: Ostergotland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Håkan Gustafsson, Adjunct Senior Lecturer, Ostergotland County Council, Sweden
Other Study IDs: NCT20210157-AI-ROL
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
Keywords: Artificial intelligence
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screened women in Region Östergötland Linkoping
  Interventions: Other: AI cancer detection system

INTERVENTIONS:
Other: AI cancer detection system — The use of AI as a third reader and as a decision support system during consensus meeting

SUMMARY:
The purpose of this observational study is to assess whether the use of AI (Transpara®) can lead to an improved quality of a double reading mammography screening program. This is investigated by performing AI as a third reader and as a decision support during the consensus meeting, compared with conventional mammography screening (double reading and consensus without AI).

DETAILED DESCRIPTION:
The AI cancer detection system will act as a 3rd reader and will recall additional cases to the consensus conference: the exams that were not recalled by double reading but are classified as the 3% most suspicious exams, based on AI derived cancer-risk scores. Secondly, AI is used as a decision support during consensus. AI risk scores and Computer-Aided Detection (CAD)-marks of suspicious calcifications and soft tissue lesions are provided to the reader(s).

The hypothesis of this study is that the use of AI has the potential to improve the quality of the screening program by increasing the cancer detection rate without affecting the recall rate.

ELIGIBILITY:
Inclusion Criteria:

* Women participating in the regular Breast Cancer Screening Program in Region Östergötland Linkoping

Exclusion Criteria:

* Women with breast implants or other foreign implants in the mammogram
* Women with symptoms or signs of suspected breast cancer

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Women eligible for population-based mammography screening
Sampling Method: Non-Probability Sample
Enrollment: 15500 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Cancer Detection rate | After 4 months of inclusion
  Proportion of women diagnosed with breast cancer among those recalled after consensus
Recall or referral rate | After 4 months of inclusion
  Proportion of women who are referred for further diagnostic workup after consensus
Positive predictive value of referrals | After 4 months of inclusion
  Proportion of women diagnosed with breast cancer among those referred

SECONDARY OUTCOMES:
Positive predictive value of Transpara® scores | After 4 months of inclusion
  Proportion of breast cancers diagnosed among women with a given AI score

CONTACTS AND LOCATIONS:
Overall Officials: Håkan Gustafsson, PhD, Principal Investigator — Linköping University - University Hospital
Locations (1):
- Region Östergötland, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rodriguez-Ruiz A, Lang K, Gubern-Merida A, Broeders M, Gennaro G, Clauser P, Helbich TH, Chevalier M, Tan T, Mertelmeier T, Wallis MG, Andersson I, Zackrisson S, Mann RM, Sechopoulos I. Stand-Alone Artificial Intelligence for Breast Cancer Detection in Mammography: Comparison With 101 Radiologists. J Natl Cancer Inst. 2019 Sep 1;111(9):916-922. doi: 10.1093/jnci/djy222. PMID 30834436
- [Background] Rodriguez-Ruiz A, Krupinski E, Mordang JJ, Schilling K, Heywang-Kobrunner SH, Sechopoulos I, Mann RM. Detection of Breast Cancer with Mammography: Effect of an Artificial Intelligence Support System. Radiology. 2019 Feb;290(2):305-314. doi: 10.1148/radiol.2018181371. Epub 2018 Nov 20. PMID 30457482
- [Background] van Winkel SL, Rodriguez-Ruiz A, Appelman L, Gubern-Merida A, Karssemeijer N, Teuwen J, Wanders AJT, Sechopoulos I, Mann RM. Impact of artificial intelligence support on accuracy and reading time in breast tomosynthesis image interpretation: a multi-reader multi-case study. Eur Radiol. 2021 Nov;31(11):8682-8691. doi: 10.1007/s00330-021-07992-w. Epub 2021 May 4. PMID 33948701
- [Background] Pinto MC, Rodriguez-Ruiz A, Pedersen K, Hofvind S, Wicklein J, Kappler S, Mann RM, Sechopoulos I. Impact of Artificial Intelligence Decision Support Using Deep Learning on Breast Cancer Screening Interpretation with Single-View Wide-Angle Digital Breast Tomosynthesis. Radiology. 2021 Sep;300(3):529-536. doi: 10.1148/radiol.2021204432. Epub 2021 Jul 6. PMID 34227882
- [Background] Raya-Povedano JL, Romero-Martin S, Elias-Cabot E, Gubern-Merida A, Rodriguez-Ruiz A, Alvarez-Benito M. AI-based Strategies to Reduce Workload in Breast Cancer Screening with Mammography and Tomosynthesis: A Retrospective Evaluation. Radiology. 2021 Jul;300(1):57-65. doi: 10.1148/radiol.2021203555. Epub 2021 May 4. PMID 33944627
- [Background] Lang K, Dustler M, Dahlblom V, Akesson A, Andersson I, Zackrisson S. Identifying normal mammograms in a large screening population using artificial intelligence. Eur Radiol. 2021 Mar;31(3):1687-1692. doi: 10.1007/s00330-020-07165-1. Epub 2020 Sep 2. PMID 32876835
- [Background] Rodriguez-Ruiz A, Lang K, Gubern-Merida A, Teuwen J, Broeders M, Gennaro G, Clauser P, Helbich TH, Chevalier M, Mertelmeier T, Wallis MG, Andersson I, Zackrisson S, Sechopoulos I, Mann RM. Can we reduce the workload of mammographic screening by automatic identification of normal exams with artificial intelligence? A feasibility study. Eur Radiol. 2019 Sep;29(9):4825-4832. doi: 10.1007/s00330-019-06186-9. Epub 2019 Apr 16. PMID 30993432
- [Background] Lang K, Hofvind S, Rodriguez-Ruiz A, Andersson I. Can artificial intelligence reduce the interval cancer rate in mammography screening? Eur Radiol. 2021 Aug;31(8):5940-5947. doi: 10.1007/s00330-021-07686-3. Epub 2021 Jan 23. PMID 33486604
- [Background] Sasaki M, Tozaki M, Rodriguez-Ruiz A, Yotsumoto D, Ichiki Y, Terawaki A, Oosako S, Sagara Y, Sagara Y. Artificial intelligence for breast cancer detection in mammography: experience of use of the ScreenPoint Medical Transpara system in 310 Japanese women. Breast Cancer. 2020 Jul;27(4):642-651. doi: 10.1007/s12282-020-01061-8. Epub 2020 Feb 12. PMID 32052311
- [Background] Kerschke L, Weigel S, Rodriguez-Ruiz A, Karssemeijer N, Heindel W. Using deep learning to assist readers during the arbitration process: a lesion-based retrospective evaluation of breast cancer screening performance. Eur Radiol. 2022 Feb;32(2):842-852. doi: 10.1007/s00330-021-08217-w. Epub 2021 Aug 12. PMID 34383147